CLINICAL TRIAL: NCT01285492
Title: A 52-week Treatment, Multi-center, Randomized, Open Label, Parallel Group Study to Assess the Long Term Safety and Tolerability of QVA149 (110 Mcg Indacaterol / 50 Mcg Glycopyrrolate o.d.) Using Tiotropium (18 Mcg o.d.) as an Active Control in Japanese Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Long Term Safety and Tolerability of QVA149 Versus Tiotropium in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQVA149A1301
Record Dates: First submitted 2011-01-25; First posted 2011-01-28 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; QVA149; NVA237; indacaterol; combination bronchodilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Tiotropium Bromide

ARMS (2):
- QVA149 (Experimental): QVA149 110/50 μg once a day (o.d)
  Interventions: Drug: QVA149
- Tiotropium (Active Comparator): tiotropium 18 μg o.d.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: QVA149 — QVA149 (110 μg indacaterol / 50 μg glycopyrronium o.d.), delivered via Concept1
  Arms: QVA149
Drug: Tiotropium — Tiotropium (18 μg o.d.), delivered via Handihaler®
  Arms: Tiotropium

SUMMARY:
This is a 52-week treatment, multi-center, randomized, open label, parallel group study to assess the long term safety and tolerability of once-daily QVA149 (indacaterol and NVA237 ([glycopyrronium bromide]) using tiotropium as an active control in Japanese patients with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe stable COPD (Stage II or Stage III) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines 2008.
* Current or ex-smokers who have a smoking history of at least 10 pack years. (Ten pack years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.)
* Patients with post-bronchodilator forced expiratory volume in one second (FEV1) ≥30% and < 80% of the predicted normal, and post-bronchodilator FEV1/forced vital capacity (FVC) < 0.7 at Visit 2.

Exclusion Criteria:

* Pregnant women or nursing mothers or women of child-bearing potential not using an acceptable method of contraception
* Patients requiring long term oxygen therapy
* Patients who have had a lower respiratory tract infection within 4 weeks prior to Visit 1
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Any patient with history of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years
* Patients with a history of certain cardiovascular comorbid conditions
* Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
* Patients in the active phase of a supervised pulmonary rehabilitation program
* Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to anticholinergic agents, long and short acting beta-2 agonists, sympathomimetic amines

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- Japan (32):
  - Novartis Investigative Site, Anjo, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Nishio, Aichi-ken
  - Novartis Investigative Site, Akita, Akita
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Kōshi, Kumamoto
  - Novartis Investigative Site, Matsusaka, Mie-ken
  - Novartis Investigative Site, Ueda, Nagano
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Kawaguhi-city, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Wakayama, Wakayama
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Ube, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 121 patients were randomized to the QVA149 group; however, demographics was on safety set and excluded 2 patients who did not take study drug
Pre-assignment Details: There was a pre-screening visit where informed consent was obtained and current COPD medications reviewed and in suitable patients, if necessary, arrangements were made to adjust prohibited COPD therapy to allowable COPD therapy. The interval between Visit 2 and 3 was a 7-days run-in period used to assess eligibility and to collect baseline values.
Groups:
- QVA149: QVA149 110/50 μg o.d. (once a day)
Period: Overall Study
Arm/Group | QVA149 | Tiotropium
Started | 121 (All patients randomized to this group) | 39 (All patients randomized to this group)
Safety Set (for Demographics) | 119 (All patients who took study drug; 2 patients did not) | 39 (All patients who took study drug)
Completed | 104 | 38
Not Completed | 17 | 1
Not completed — Adverse Event | 11 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | Tiotropium | Total
Number analyzed (Participants) | 119 | 39 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (6.79) | 69.4 (6.90) | 69.3 (6.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 114 | 37 | 151
Baseline Weight [Mean (Standard Deviation); unit: kg] | 60.38 (9.613) | 61.44 (8.788) | 60.64 (9.400)
Baseline Height [Mean (Standard Deviation); unit: cm] | 164.4 (7.08) | 163.3 (6.38) | 164.1 (6.91)
Baseline Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.31 (3.067) | 23.02 (2.919) | 22.49 (3.037)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) or Death
Description: An AE was the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event was not considered to be related to study drug. Study drug includes the investigational drug under evaluation and the comparator drug or placebo that was given during any phase of the study. Adverse events starting on or after the time of the first inhalation of study drug were classified as a treatment emergent adverse event.
Time Frame: 52 weeks
Population: The safety set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Participants
  Adverse Events (AEs) | 101 | 28
  Serious Advers Events (SAEs) | 19 | 2
  Death | 1 | 0

2. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Hematology Values at Any Timepoint Over the Whole Treatment Period
Description: Clinically notable hematology values were: hemoglobin - male <11.5g/dL, female <9.5 g/dL; hematocrit - male <37%, female <32%; white cell count - <2800µL or >16000µL; platelets - <7.5 10*4/µL or >70.0 10*4/µL
Time Frame: 52 weeks
Population: The safety set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Participants
  Hemoglobin: male (n = 113, 36) | 3 | 0
  Hemoglobin: female (n = 5, 2) | 0 | 0
  Hematocrit: male (n = 113, 36) | 6 | 0
  Hematocrit: female (n = 5, 2) | 0 | 0
  White Cell Count < 2800 (n = 118, 38) | 0 | 0
  White Cell Count > 2800 (n = 118, 38) | 0 | 0
  Platelets < 7.5 (n = 118, 38) | 0 | 0
  Platelets > 70.0 (n = 118, 38) | 0 | 0

3. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Biochemistry Values at Any Time-point Over the Treatment Period
Description: Clinically notable biochemistry values were: total protein - <4.0 g/dL or >9.5 g/dL; albumin <2.5 g/dL; bilirubin (total) >1.9 mg/dL; BUN >27 mg/dL; creatinine >1.99 mg/dL; AST >3 x ULN U/L; ALT >3 x ULN U/L; ALP >3 x ULN U/L; y-GTP >3 x ULN U/L; sodium <125 mEq/L or >160 mEq/L; potassium <3.0 mEq/L or >6.0 mEq/L; glucose <51.0 mg/dL or >180.0 mg/dL
Time Frame: 52 weeks
Population: The safety set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Participants
  Total protein - <4.0 g/dL (n = 118, 38) | 0 | 0
  Total protein - > 9.5 g/dL (n = 118, 38) | 0 | 0
  albumin <2.5 g/dL (n = 118, 38) | 0 | 0
  bilirubin (total) >1.9 mg/dL (n = 118, 38) | 0 | 0
  BUN >27 mg/dL (n = 118, 38) | 1 | 0
  creatinine >1.99 mg/dL (n = 118, 38) | 0 | 0
  AST >3 x ULN U/L (n = 118, 38) | 0 | 0
  ALT >3 x ULN U/L (n = 118, 38) | 0 | 0
  ALP >3 x ULN U/L (n = 118, 38) | 0 | 0
  y-GTP >3 x ULN (n = 118, 38) | 2 | 2
  sodium <125 mEq/L (n = 118, 38) | 0 | 0
  sodium >160 mEq/L (n = 118, 38) | 0 | 0
  potassium <3.0 mEq/ (n = 118, 38) | 0 | 0
  potassium >6.0 mEq/ (n = 118, 38) | 0 | 0
  glucose <51.0 mg/dL (n = 118, 38) | 0 | 0
  glucose >180.0 mg/dL (n = 118, 38) | 7 | 3

4. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Vital Signs Values at Any Time-point Over the Whole Treatment Period
Description: Clinically notable vital sign values were: pulse rate - low, <40 bpm or <=50 bpm and decrease from baseline >=15bpm; pulse rate high, >130 bpm or >=120bpm and increase from baseline >=15 bpm. Systolic blood pressure - low, <75 mmHg or <=90 mmHg and decrease from baseline >=20 mmHg; high, >200 mmHg or >=180 mmHg and increase from baseline >=20 mmHg. Diastolic blood pressure - low, <40 mmHg or <=50 mmHg and decrease from baseline >=15 mmHg; high, >115 mmHg or >=105 mmHg and increase from baseline >=15 mmHg.
Time Frame: 52 weeks
Population: The safety set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Participants
  Pulse rate: low | 0 | 0
  Pulse rate: high | 0 | 0
  Pulse rate: low or high | 0 | 0
  Systolic blood pressure - low | 4 | 0
  Systolic blood pressure - high | 0 | 1
  Systolic blood pressure - low or high | 4 | 1
  Diastolic blood pressure - low | 3 | 0
  Diastolic blood pressure - high | 2 | 1
  Diastolic blood pressure - low or high | 5 | 1

5. Secondary Outcome: Number of Patients With Newly Occurring or Worsening Clinically Notable Fridericia's QTc Values at Any Time-point Over the Whole Treatment Period
Description: Clinically notable change from baseline was an increase from baseline of 30 or greater milliseconds (ms).
Time Frame: 52 weeks
Population: The safety set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Participants
  Males: QTc > 450 ms (n = 111, 36) | 6 | 0
  Females: QTc > 470 ms (n = 5, 2) | 0 | 0
  Increase from baseline 30 to 60 ms (n = 116, 38) | 12 | 3
  Increase from baseline > 60 ms (n = 116, 38) | 1 | 0

6. Secondary Outcome: Change in Pre-dose Forced Expiratory Volume in One Second (FEV1) From Baseline
Description: Pre-dose FEV1 is defined as the average of the measurements at 45 and 15 min pre-dose. Baseline is defined as the pre-dose FEV1 value on Day 1 (Week 1).
Time Frame: Weeks 3, 6, 12, 24, 36, 52
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Litres
  Week 3 (117, 38) | 0.206 (0.1534) | 0.093 (0.0977)
  Week 6 (115, 38) | 0.202 (0.1668) | 0.083 (0.1201)
  Week 12 (113, 38) | 0.209 (0.1725) | 0.139 (0.1562)
  Week 24 (113, 37) | 0.198 (0.1735) | 0.115 (0.1400)
  Week 36 (105, 37) | 0.182 (0.1619) | 0.082 (0.1465)
  Week 52 (104, 37) | 0.189 (0.1762) | 0.052 (0.1688)

7. Secondary Outcome: Change in Pre-dose Forced Vital Capacity (FVC) From Baseline
Description: Pre-dose FVC is defined as the average of the measurements at 45 and 15 min pre-dose. Baseline is defined as the pre-dose FVC value on Day 1 (Week 1).
Time Frame: Weeks 3, 6, 12, 24, 36, 52
Population: Full Analysis Set (FAS) included all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | QVA149 | Tiotropium
Number analyzed (Participants) | 119 | 39
Litres
  Week 3 (117, 38) | 0.314 (0.2882) | 0.213 (0.2369)
  Week 6 (115, 38) | 0.310 (0.3178) | 0.173 (0.2162)
  Week 12 (113, 38) | 0.335 (0.2948) | 0.279 (0.2942)
  Week 24 (113, 37) | 0.330 (0.3248) | 0.206 (0.2367)
  Week 36 (105, 37) | 0.264 (0.2706) | 0.167 (0.2438)
  Week 52 (104, 37) | 0.261 (0.3047) | 0.112 (0.2462)

ADVERSE EVENTS:
Arm/Group | QVA149 | Tiotropium
Serious Adverse Events (participants affected / at risk) | 19/119 | 2/39
Other Adverse Events (participants affected / at risk) | 66/119 | 23/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=119) | Tiotropium (N=39)
Arrhythmogenic right ventricular dysplasia (Congenital, familial and genetic disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 3 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=119) | Tiotropium (N=39)
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 3
Influenza (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 40 | 12
Pharyngitis (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 6
Rib fracture (Injury, poisoning and procedural complications) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Headache (Nervous system disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 4 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 29 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.